CLINICAL TRIAL: NCT00040183
Title: A Randomized Placebo Controlled Study of OSI-774 (Tarceva (TM)) Plus Gemcitabine in Patients With Locally Advanced, Unresectable or Metastatic Pancreatic Cancer
Brief Title: OSI-774 (Tarceva) Plus Gemcitabine in Patients With Locally Advanced, Unresectable or Metastatic Pancreatic Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA.3
Record Dates: First submitted 2002-06-21; First posted 2002-06-25 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2015-06

CONDITIONS: Pancreatic Cancer
Keywords: Tarceva, EGFR, erlotinib, OSI-774
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Tarceva (erlotinib HCl, OSI-774)

SUMMARY:
The purpose of this study is to determine if OSI-774 will improve overall survival when combined with a standard dose of the chemotherapy drug gemcitabine, to individuals with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed diagnosis of adenocarcinoma of the pancreas;cancer which is unresectable, locally advanced or metastatic.

Must have evidence of disease (clinical or radiological). Male or female, 18 years or older. Patients may have received prior radiation treatment for management of local disease providing that disease progression has been documented.

All toxicities have resolved, and the last fraction of radiation treatment was completed at least 4 weeks prior to randomization.

Patients may not have received prior chemotherapy, other then 5FU (+/- folic acid) or gemcitabine given concurrently with radiation treatment as a 'radiosensitiser.'

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2001-11-29 (Actual); Primary Completion 2004-01-15 (Actual); Study Completion 2004-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (140):
- United States (60):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Loma Linda University Cancer Institute, Loma Linda, California
  - Metropolitan Hematology/Oncology Medical Group, Inc., Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Kaiser Permanente, San Diego, California
  - DeQuattro Community Cancer Center, Manchester, Connecticut
  - New Britain General Hospital, New Britain, Connecticut
  - Eastern Connecticut Oncology, Norwich, Connecticut
  - Carl and Dorothy Bennett Cancer Center, Stamford, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Oncology Hematology Group of South Florida, Miami, Florida
  - Ocala Oncology, Ocala, Florida
  - Tampa General Hospital, Tampa, Florida
  - Atlanta Cancer Center, Atlanta, Georgia
  - Onc/Hem Associates of Central Illinois, Peoria, Illinois
  - Hematology Oncology Associates of Illinois, Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - University of Iowa Hospital & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Norton Healthcare, Inc., Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - J Gurtler, Hematology and Oncology, Metairie, Louisiana
  - Annapolis Medical Specialists, Annapolis, Maryland
  - Sinai Hospital, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - St Elizabeth Medical Center, Boston, Massachusetts
  - New England Medical Center, Boston, Massachusetts
  - Berkshire Hematology & Oncology, PC, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri
  - New Hampshire Oncology-Hematology PA, Hooksett, New Hampshire
  - St Barnabas Medical Center, Livingston, New Jersey
  - Arena Oncology Associates, Great Neck, New York
  - New York University School of Medicine, New York, New York
  - St Luke's-Roosevelt Hospital, New York, New York
  - Interlakes Oncology & Hematology, P.C., Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Odyssey Research Services, Bismarck, North Dakota
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Chiles Research Cancer Center, Portland, Oregon
  - Hematology & Oncolgy Assoc of NE PA, Dunmore, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Charleston Hematology/Oncology, Charleston, South Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Arlington Cancer Centre, Arlington, Texas
  - Southwest Regional Cancer Center, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Tyler Hematology Oncology PA, Tyler, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Hematology & Oncology Associates of Virginia, Ltd., Richmond, Virginia
  - Western Washington Oncology Inc., Olympia, Washington
  - Southwest Washington Medical Center, Vancouver, Washington
  - Oncology of Wisconsin, Milwaukee, Wisconsin
- Argentina (6):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Britanico, Buenos Aires
  - Instituto Oncologico Angel Roffo, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Hospital Churruca Visca, Buenos Aires
  - Centro Medico Confidence, Buenos Aires
- Australia (8):
  - Concord Hospital, Concord, New South Wales
  - Newcastle Mater Hospital, HRMC Waratah, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Ashford Cancer Centre, Ashford, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Frankston Hospital, Frankston, Victoria
  - Austin & Repatriation Medical Centre, Heidelberg, Victoria
- Institute Jules Bordet, Brussels, Belgium
- Brazil (4):
  - Nucleo de Oncolgia da Bahia, Salvador, Estado de Bahia
  - Hospital Vera Cruz S/A, Barro Prêto, Minas Gerais
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
- Canada (25):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - Pentincton Regional Hospital, Pentincton, British Columbia
  - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA VAncouver Centre, Vancouver, British Columbia
  - BCCA- Vancouver Island Centre, Victoria, British Columbia
  - CancerCare Manitoba (CCMB), Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - London Regional Cancer Center, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Group Health Centre, Saulte Ste. Marie, Ontario
  - Hotel Dieu Health Sciences HospitalNiagra, St. Catharines, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto-Sunnybrook Regional Cancer Center, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - St Joseph's Health Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hopital Du Sacre-Coeur, Montreal, Quebec
  - Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Clinica Las Condes, Las Condes, Chile
- Germany (7):
  - Charite Campus Virchow Klinikum, Berlin
  - Universitatsklinikum Essen, Essen
  - Tumor Biology Center, Freiburg im Breisgau
  - Universitatskliniken des Saarlands Innere Medizin II, Hamburg
  - Innere MedizinUniversitatsklinikum Heidelberg, Heidelberg
  - Universitatskliniken des Saarlands, Homburg
  - Medizinische Poliklinik der Universitaet Wurzburg, Würzburg
- Greece (2):
  - Anticancer Hospital of Thessaloniki "THEAGENIO", Thessaloniki
  - District General Hospital of Thessaloniki "HIPPOKRATION", Thessaloniki
- Israel (5):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center (Belinson Campus), Petach Tiqva
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center (Ichikov), Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Azienda Ospedaliera Universitaria Policlinico A.O.V.P. Oncologia Medica, Palermo, Italy
- Instituto Nacional De Cancerologia, Mexico City, Mexico
- New Zealand (2):
  - Auckland Hospital, Auckland
  - Christchurch HospitalClinical Oncology Hospital, Christchurch
- Poland (2):
  - Great Poland Cancer Centre, Poznan
  - Dolnoslaskie Centrum Onkologii, Wroclaw
- Romania (3):
  - Oncology Institute Ion Chiricuta, Cluj-Napoca
  - St. Spiridon University Hospital, Iași
  - Clinical County Hospital Sibiu, Sibiu
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Cancer Centre, Singapore
- United Kingdom (9):
  - ICRF Medical Oncology Unit, Oxford, Oxfordshire
  - Velindre Hospital, Cardiff, Wales
  - Russell's Hall HospitalDepartment of OncologyGeorgina Unit, Dudley, West Midlands
  - Deanesly Centre, Wolverhampton, West Midlands
  - The Princess Royal Hospital, Hull
  - St. Bartholomews Hospital, London
  - North Middlesex Hospital, London
  - Department of Medical Oncology, Manchester
  - Newcastle General Hospital, Newcastle upon Tyne

REFERENCES:
- [Background] Moore MJ, Goldstein D, Hamm J, Figer A, Hecht JR, Gallinger S, Au HJ, Murawa P, Walde D, Wolff RA, Campos D, Lim R, Ding K, Clark G, Voskoglou-Nomikos T, Ptasynski M, Parulekar W; National Cancer Institute of Canada Clinical Trials Group. Erlotinib plus gemcitabine compared with gemcitabine alone in patients with advanced pancreatic cancer: a phase III trial of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 May 20;25(15):1960-6. doi: 10.1200/JCO.2006.07.9525. Epub 2007 Apr 23. PMID 17452677
- [Derived] Shultz DB, Pai J, Chiu W, Ng K, Hellendag MG, Heestand G, Chang DT, Tu D, Moore MJ, Parulekar WR, Koong AC. A Novel Biomarker Panel Examining Response to Gemcitabine with or without Erlotinib for Pancreatic Cancer Therapy in NCIC Clinical Trials Group PA.3. PLoS One. 2016 Jan 25;11(1):e0147995. doi: 10.1371/journal.pone.0147995. eCollection 2016. PMID 26808546
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=62